CLINICAL TRIAL: NCT04383977
Title: A Phase 2 Randomized, Open-label, Multicenter Trial of Apatinib and Etoposide Capsule Versus Apatinib in Patients With Platinum Resistant or Refractory Ovarian Cancer
Brief Title: Apatinib and Etoposide Capsule Versus Apatinib in Patients With Platinum Resistant Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-OC-203
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib-Etoposide capsule (Experimental): Apatinib (375 mg qd, q3w) and Etoposide capsule(50 mg/d, d1-14, q3w) combination until disease progression or intolerable toxicity
  Interventions: Drug: Apatinib and Etoposide capsule
- Apatinib (Active Comparator): Apatinib (375 mg qd, q3w) until disease progression or intolerable toxicity
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib and Etoposide capsule — Apatinib (375 mg qd, q3w) and Etoposide capsule(50 mg/d, d1-14, q3w) combination until disease progression or intolerable toxicity
  Arms: Apatinib-Etoposide capsule
Drug: Apatinib — Apatinib (375 mg qd, q3w) until disease progression or intolerable toxicity
  Arms: Apatinib

SUMMARY:
The study is conducted to evaluate the efficacy, safety and tolerability of apatinib (375 mg qd) or apatinib (375 mg qd) and etoposide capsule (50 mg/d, d1-14, q3w) in subjects with platinum resistant or refractory ovarian cancer compared with apatinib (375 mg qd).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, ≥18 Years.
2. Epithelial ovarian, fallopian tube or primary peritoneal cancer
3. Platinum refractory and resistant disease (disease progression during platinum therapy or within <6 months of platinum therapy)
4. EOCG performance status of 0-2

Exclusion Criteria:

1. Non-epithelial tumours
2. Ovarian tumours with low malignant potential
3. Surgery (including open biopsy) within 4 weeks before starting study therapy or anticipated need for major surgery during study treatment
4. Evidence of rectosigmoid involvement by pelvic examination, bowel involvement on computed tomography, or clinical symptoms of bowel obstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by investigator | up to 2 years
  ORR was defined as the proportion of subjects who have a complete or partial response relative to baseline .

SECONDARY OUTCOMES:
AEs+SAEs | 30 days after the last dose
  Frequency and severity of Adverse Events or Serious Adverse Events as defined by CTCAE version 5.0
PFS by investigator | up to 2 years
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigator according to the RECIST criteria.
Overall Survival (OS) | up to 3 years
  OS is the time interval from the date of randomization to death from any cause.
Pharmacokinetic characteristic | up to 2 years
  Evaluation of PK parameters Tmax of apatinib or etoposide in plasma
Pharmacokinetic characteristic | up to 2 years
  Evaluation of PK parameters Cmax of apatinib or etoposide in plasma
Pharmacokinetic characteristic | up to 2 years
  Evaluation of PK parameters t1/2 of apatinib or etoposide in plasma
Pharmacokinetic characteristic | up to 2 years
  Evaluation of PK parameters AUC0-t of apatinib or etoposide in plasma

IPD SHARING:
Plan to Share IPD: No
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

REFERENCES:
- [Derived] Hou Z, Lan C, Huang X, Salcedo-Hernandez RA, El-Tawab S. Efficacy, safety and pharmacokinetics of apatinib plus etoposide versus apatinib alone for platinum-resistant recurrent ovarian cancer: protocol of a multicenter, open-label, randomized phase 2 trial. Transl Cancer Res. 2023 Oct 31;12(10):2959-2967. doi: 10.21037/tcr-23-1924. Epub 2023 Oct 26. PMID 37969395
- See also: ClinicalTrials.gov Results Data Element Definitions for Interventional and Observational Studies — https://prsinfo.clinicaltrials.gov/results_definitions.html
- See also: Checklists, templates, and examples to help gather information needed to report results to ClinicalTrials.gov — https://prsinfo.clinicaltrials.gov/results_table_layout/ResultSimpleForms.html